CLINICAL TRIAL: NCT05060055
Title: Volumetric Digital Analysis on the Effect of a Customized Healing Abutment With or Without Connective Tissue Graft at Maxillary Immediate Implant Sites - A Randomized Clinical Trial
Brief Title: Digital Assessment at Peri-implant Tissues After Immediate Implants With Customized Healing Abutments and Connective Tissue Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Católica Portuguesa (Other)
Responsible Party: Principal Investigator, Tiago Borges, Adjunct-Professor, Head of Oral Surgery, Center for Interdisciplinary Research in Health. Faculty of Dental Medicine, Universidade Católica Portuguesa, Viseu, Portugal., Universidade Católica Portuguesa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCatolicaPortuguesa
Record Dates: First submitted 2021-07-26; First posted 2021-09-28 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Dental Implant Failed
Keywords: autografts; wound healing; three-dimensional imaging; treatment outcome; dental implants; alveolar ridge augmentation; alveolar bone loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: The present study was designed as a prospective, controlled clinical trial with a parallel-group design and balanced randomization (ratio 1:1)
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Customized healing abutment inserted in immediate implant placement in association with the use of a connective tissue graft.
  Interventions: Procedure: Immediate dental implant placement
- Control Group (Active Comparator): Customized healing abutment inserted in immediate implant placement.
  Interventions: Procedure: Immediate dental implant placement

INTERVENTIONS:
Procedure: Immediate dental implant placement — Immediate dental implant placement

SUMMARY:
After a single-tooth extraction, physiological remodeling processes are unavoidable which leads to a total loss of the periodontal ligament and resorption of the bundle bone. Immediate implant placement associated with bone substitutes and customized healing abutments seems to reduce the amount of resorption at peri-implant areas. Recently, studies evaluating the use of a connective tissue grafts are being conducted in order to assess possible final outcome advantages in immediate implant procedures. This study aims to evaluate peri-implant tissue dimensional changes after the use of a customized healing abutment with or without connective tissue graft in flapless maxillary immediate implant placement.

DETAILED DESCRIPTION:
The present study was designed as a prospective, controlled clinical trial with a parallel-group design and balanced randomization (ratio 1:1) to document the peri-implant tissues response in using a customized healing abutment with a connective tissue graft (Test group) or without a connective tissue graft (Control group) xenogeneic collagen matrix (Group CM) or a customized healing abutment (Group CA) in flapless maxillary immediate implants. The protocol was reviewed and approved by the Institute of Bioethics of the Catholic University of Portugal (Project nº 139) and the patients included will be previously informed to participate in this investigation signing an informed consent considering the 1975 Declaration of Helsinki, revised in 2013. Group designation will be kept in opaque-sealed envelopes that will be opened after implant insertion by an investigator (D.F), not involved in surgical procedures, randomly allocating participants to one of the two treatment groups. Patients' inclusion criteria are: 1) ≥18 years of age; 2) patients who had a failing tooth and needed an implant placing therapy in the aesthetic zone (between 15-25); 3) the failing tooth has adjacent and opposing natural teeth; 4) sufficient mesial-distal and inter-occlusal space for placement of the implant and definitive restoration; 5) had an intact socket wall previously to the extraction; 6) had sufficient apical bone to place an immediate implant with minimum primary stability of 30 N/cm. Exclusion criteria are: individuals diagnosed with periodontal disease; medical and general contraindications for the surgical procedure; heavy smokers (> 10 cigarettes/day); an active infection at the implant site. A CONSORT 2010 check-list will be also performed in order to consider an appropriate guideline for the present randomized trial study.

All surgical procedures will be conducted under appropriate local anesthesia 4% articaine with adrenaline 1:100000 (UbistesinTM, 3M-ESPE, St. Paul, MN, USA). In both groups, flapless tooth extractions will be performed after sectioning the tooth, followed by the use of periotomes and elevators to separate the two parts of the tooth, avoiding damage to the buccal and palatal bone plates. All patients will be treated with cylindrical shape implants (OsseoSpeed EV™, AstraTech Implant System, Dentsply Implants, Möhndal, Sweden) with a narrow diameter internal connection platform following the surgical sequence protocol provided by the manufacturer. Both groups will receive a customized healing abutment made of polymethyl methacrylate (PMMA) material, designed and fabricated accordingly with the gingival contour of the original tooth. Patients included in the Test group will receive connective tissue grafts harvested using the single incision technique.

A protocol was elaborated to study the variables of interest. One examiner, blinded for the surgical procedure, will be calibrated through an intra-examiner test (Dahlberg d-value), consisting in a double consecutive data collection of 10 randomly chosen patients included in this study.

Data collection will be performed in four appointments. A Cone Beam Computer Tomography (CBCT) evaluation (Ortophos XG 3D®, Sirona Dental Systems GmbH, Bensheim, Germany) will be performed before tooth extraction and implant placement (T0). At this point, two clinical parameters will be assessed with a periodontal probe (PCB 12; Hu-Friedy, Chicago, IL, USA) to the nearest millimeter: BID (distance between implant shoulder and the buccal bone plate) and KM (distance between the gingival groove and the mucogingival junction). Digital impressions (Cerec Omnicam®, Sirona Dental Systems GmbH, Bensheim, Germany) will be taken prior to extraction (T0), one month (T1), four months (T2) and 12 months (T3) after implant insertion allowing to superimpose the digital files and to evaluate volumetric changes between different time points at peri-implant tissue areas like Buccal Volume Variation (BVv) and Total Volume Variation (TVv). Mucosa variation between T0 and T3 will be digitally computed assessing the papilla presence at mesial (MPHv) and distal (DPHv) sites and the mucosa height (MGHv). Mean values will be compared and statistical significance will be at 0,05.

ELIGIBILITY:
Inclusion Criteria:

* 1) ≥18 years of age; 2) patients who had a failing tooth and needed an implant placing therapy in the aesthetic zone (between 15-25); 3) the failing tooth has adjacent and opposing natural teeth; 4) sufficient mesial-distal and inter-occlusal space for placement of the implant and definitive restoration; 5) had an intact socket wall previously to the extraction; 6) had sufficient apical bone to place an immediate implant with minimum primary stability of 30 N/cm.

Exclusion Criteria:

* individuals diagnosed with periodontal disease; medical and general contraindications for the surgical procedure; heavy smokers (> 10 cigarettes/day); an active infection at the implant site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Buccal volume variation (BVvT0) | Baseline (T0); 1 month (T1); 4 months (T2) and 12 months (T3)
  Variation of the alveolar volume at the buccal aspect. The 3D-analysis was conducted with "Boolean" functions, which allowed researchers to obtain the volume variation in each time point from different variables like the Buccal Volume Variation (BVv0-1, BVv0-2, and BVv0-3), computed in cubic millimetres (mm3) and To allow a direct comparison of different sites at different time points, relative percentages of these variables were calculated based on the ROI volume at T0.
Buccal volume variation (BVvT1) | 1 month (T1)
  Variation of the alveolar volume at the buccal aspect. The 3D-analysis was conducted with "Boolean" functions, which allowed researchers to obtain the volume variation in each time point from different variables like the Buccal Volume Variation (BVv0-1, BVv0-2, and BVv0-3), computed in cubic millimetres (mm3) and To allow a direct comparison of different sites at different time points, relative percentages of these variables were calculated based on the ROI volume at T0.
Buccal volume variation (BVvT2) | 4 months (T2)
  Variation of the alveolar volume at the buccal aspect. The 3D-analysis was conducted with "Boolean" functions, which allowed researchers to obtain the volume variation in each time point from different variables like the Buccal Volume Variation (BVv0-1, BVv0-2, and BVv0-3), computed in cubic millimetres (mm3) and To allow a direct comparison of different sites at different time points, relative percentages of these variables were calculated based on the ROI volume at T0.
Buccal volume variation (BVvT3) | 12 months (T3)
  Variation of the alveolar volume at the buccal aspect. The 3D-analysis was conducted with "Boolean" functions, which allowed researchers to obtain the volume variation in each time point from different variables like the Buccal Volume Variation (BVv0-1, BVv0-2, and BVv0-3), computed in cubic millimetres (mm3) and To allow a direct comparison of different sites at different time points, relative percentages of these variables were calculated based on the ROI volume at T0.
Total volume variation (TVvT0) | Baseline (T0); 1 month (T1); 4 months (T2) and 12 months (T3)
  Variation of the alveolar volume at the buccal and palatal side. The 3D-analysis was conducted with "Boolean" functions, which allowed researchers to obtain the volume variation in each time point from different variables like the Total Volume Variation (TVv0-1, TVv0-2, e TVv0-3), computed in cubic millimetres (mm3) and To allow a direct comparison of different sites at different time points, relative percentages of these variables were calculated based on the ROI volume at T0
Total volume variation (TVvT0) | Baseline (T0)
  Variation of the alveolar volume at the buccal and palatal side. The 3D-analysis was conducted with "Boolean" functions, which allowed researchers to obtain the volume variation in each time point from different variables like the Total Volume Variation (TVv0-1, TVv0-2, e TVv0-3), computed in cubic millimetres (mm3) and To allow a direct comparison of different sites at different time points, relative percentages of these variables were calculated based on the ROI volume at T0
Total volume variation (TVvT1) | 1 month (T1)
  Variation of the alveolar volume at the buccal and palatal side. The 3D-analysis was conducted with "Boolean" functions, which allowed researchers to obtain the volume variation in each time point from different variables like the Total Volume Variation (TVv0-1, TVv0-2, e TVv0-3), computed in cubic millimetres (mm3) and To allow a direct comparison of different sites at different time points, relative percentages of these variables were calculated based on the ROI volume at T0
Total volume variation (TVvT2) | 4 months (T2)
  Variation of the alveolar volume at the buccal and palatal side. The 3D-analysis was conducted with "Boolean" functions, which allowed researchers to obtain the volume variation in each time point from different variables like the Total Volume Variation (TVv0-1, TVv0-2, e TVv0-3), computed in cubic millimetres (mm3) and To allow a direct comparison of different sites at different time points, relative percentages of these variables were calculated based on the ROI volume at T0
Total volume variation (TVvT3) | 12 months (T3)
  Variation of the alveolar volume at the buccal and palatal side. The 3D-analysis was conducted with "Boolean" functions, which allowed researchers to obtain the volume variation in each time point from different variables like the Total Volume Variation (TVv0-1, TVv0-2, e TVv0-3), computed in cubic millimetres (mm3) and To allow a direct comparison of different sites at different time points, relative percentages of these variables were calculated based on the ROI volume at T0

SECONDARY OUTCOMES:
Buccal wall thickness (BT) | Baseline
  measurement of the facial bone wall. The acquisition of radiographic images was performed with a volumetric dimension of 8 x 8 cm for 14s with the XG 3D tomography acquisition protocol, with a voxel size of 0.1 mm in HD mode. BT was measured 1 mm above the coronal bone margin using a central slice, as well at the mesial and distal slices, ranging 1 mm from the central slice. Mean BT values were obtained as the average values of the three slices. Measurements were made in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Católica Portuguesa, Viseu, Portugal

REFERENCES:
- [Derived] Fernandes D, Marques T, Borges T, Montero J. Volumetric analysis on the use of customized healing abutments with or without connective tissue graft at flapless maxillary immediate implant placement: A randomized clinical trial. Clin Oral Implants Res. 2023 Sep;34(9):934-946. doi: 10.1111/clr.14119. Epub 2023 Jun 29. PMID 37386752

DOCUMENTS (1):
  • Informed Consent Form (2021-04-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT05060055/ICF_000.pdf